CLINICAL TRIAL: NCT06062901
Title: Survivorship ECHO Project
Brief Title: An Educational Intervention on Provider Knowledge for the Support of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Ashley Davenport, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-21149; NCI-2021-06471 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-09-12; First posted 2023-10-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (Survivorship ECHO) (Experimental): Participants attend 6 sessions of Survivorship ECHO educational intervention over 1 hour each, every 2 weeks for 12 weeks. Participants may optionally participate in a one-on-one interview to give feedback about the sessions over 30 minutes.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational intervention
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Interview — Participate in one-on-one interview
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial utilizes the Project Extension for Community Healthcare Outcomes (ECHO) model to recruit, train, and support community healthcare providers in cancer survivorship best practices. Cancer survivors have distinct medical needs and are more likely to report being in poor or fair overall health compared to those who do not report a history of cancer. There is a lack of educational opportunities focused on survivorship care for health providers. Although progress has been made with the development of survivorship guidelines, physicians continue to express barriers to addressing concerns of cancer survivors. This study is to utilize a Survivorship ECHO education intervention to assess its effects on provider knowledge and comfort with survivorship guidelines as well as greater adherence to guideline concordant breast cancer survivorship care recommendations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effectiveness of the Survivorship ECHO's platform by assessing provider knowledge of cancer survivorship best practices using pre- and post-enrollment surveys.

II. Evaluate implementation of survivorship best practices into clinical practice and documentation after enrollment in our Survivorship ECHO.

OUTLINE:

Participants attend 6 sessions of Survivorship ECHO educational intervention over 1 hour each, every 2 weeks for 12 weeks. Participants may optionally participate in a one-on-one interview to give feedback about the sessions over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Providers from The James Cancer Network (consists of five community sites in Ohio: St. Rita's Memorial Center, Memorial Health, Madison Health, Wooster Community Hospital, and Clinton Memorial Hospital)
* Eligible participants will include registered nurses, advanced practice registered nurses, physician assistants, nutritionists, radiation oncologists and oncologists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in level of understanding in key survivorship knowledge areas | Baseline up to study completion, typically 1 year
  Includes knowledge on surveillance, late and long-term effects of chemotherapy, health promotion, disease prevention and psychosocial evaluation and support. A Likert survey will assess provider comfort and knowledge with core cancer survivorship competencies with higher scores associated with higher levels of knowledge and comfort.
Met and unmet needs | Up to study completion, typically 1 year
  Content, participant needs, and aspects of delivering the Survivorship ECHO platform explored using qualitative analysis.
Acceptability of current structure | Up to study completion, typically 1 year
  Content, participant needs, and aspects of delivering the Survivorship ECHO platform explored using qualitative analysis.
Barriers to accessing ECHO | Up to study completion, typically 1 year
  Content, participant needs, and aspects of delivering the Survivorship ECHO platform explored using qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Davenport, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT06062901/ICF_001.pdf